CLINICAL TRIAL: NCT05816512
Title: Antimicrobial Efficacy of Biogenic Gold Nano Particle From Pelargonium Graveolens Leaves Extract Mouthwash for Children. (A Randomized Controlled Trial)
Brief Title: Antimicrobial Efficacy of Biogenic Gold Nano Particle From Pelargonium Graveolens Leaves Extract Mouthwash for Children
Acronym: GNPG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahmed Yousif Mahdi (Other)
Collaborators: University of Baghdad (Other)
Responsible Party: Sponsor-Investigator, Ahmed Yousif Mahdi, Principal Investigator, University of Baghdad
Organization: University of Baghdad (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Antimicrobial Mouthwash
Record Dates: First submitted 2023-03-31; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Dental Caries; Gingivitis; Periodontitis
Keywords: Dental caries Gold Nanoparticle Pelargonium Graveolens
MeSH Terms: conditions — Dental Caries; Gingivitis; Periodontitis | interventions — chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Single (participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gold Nano particle from Pelargonium Graveolens Mouthwash group (Experimental): Gold Nano particle from Pelargonium Graveolens Mouthwash will be applied as a mouthwash for three weeks and then follow up .
  Interventions: Drug: Gold Nano particle from Pelargonium Graveolens Mouthwash
- Chlorhexidine gluconate mouth wash group (Active Comparator): Chlorhexidine gluconate mouth wash will be applied as a mouthwash for three weeks and then follow up .
  Interventions: Drug: Chlorhexidine gluconate mouthwash .

INTERVENTIONS:
Drug: Gold Nano particle from Pelargonium Graveolens Mouthwash — Gold Nano particle from Pelargonium Graveolens Mouthwash will be applied by using 15ml of it for one minute, two times daily for three weeks and then follow up after three weeks the clinical parameters as ( plaque index, gingival index and calculus index ) and microbiological aspect will be assessed .
  Other Names: Gold Nano particle Pelargonium Graveolens
  Arms: Gold Nano particle from Pelargonium Graveolens Mouthwash group
Drug: Chlorhexidine gluconate mouthwash . — Chlorhexidine gluconate mouthwash will be applied by using 15ml of it for one minute, two times daily for three weeks and then follow up after three weeks the clinical parameters as ( plaque index, gingival index and calculus index ) and microbiological aspect will be assessed .
  Other Names: Chlorhexidine gluconate
  Arms: Chlorhexidine gluconate mouth wash group

SUMMARY:
The study is randomized controlled trial ... The null hypothesis of the present study is that there is no antibacterial efficacy of gold nanoparticles of pelargonium graveolens mouthwash against Streptococcus mutans and Candida Albicans . Meanwhile the alternative hypothesis of the present study is that gold nanoparticles of pelargonium graveolens mouthwash have antimicrobial activity against Streptococcus mutans and Candida Albicans .

DETAILED DESCRIPTION:
This is double blind study will be conducted among male patients with mild to moderate gingivitis . Those patients aged between (7-14 ) years old who attended the second specialized dental health center in Baquba city/ Diyala governorate/ Iraq. patients will be randomly assigned to one of two study groups the first group is Gold Nano particle from Pelargonium Graveolens Mouthwash , the second Chlorhexidine. by using 15ml of it for one minute two times daily for three weeks. In this study a clinical parameters as ( plaque index, gingival index and calculus index ) were assessed at the base line (before mouthwash use), and then assessed three times at one week interval after the base line assessment through the period of mouthwash use. On the other hand, microbiological aspect were assessed for those patients before and three weeks after the use of Gold Nano particle from Pelargonium Graveolens Mouthwash and Chlorhexidine . After three weeks the mean of plaque, gingival, and culculs indices are significantly reduced after the use of Biogenic Gold Nano particle from Pelargonium Graveolens Leaves Extract Mouthwash.

ELIGIBILITY:
Inclusion Criteria:

* The study sample will include a group if children aged (7-14) years, with mild to moderate crowding, attending the specialist dental center in Diyala city.
* Patients with mild to moderate gingivitis as a base line (for standardization).
* Healthy child without any oral ulceration or systemic medical condition.
* Cooperative child.
* Patient did not take any antibiotics or anti-fungal for at least 4 weeks prior to sampling procedure.
* Children are healthy without any systemic disease .
* From the same geographical area ( Diyala Governorate ).

Exclusion Criteria:

* Children outside specified age.
* Children with systemic disease or on medication.
* Children on a daily fluoride or other therapeutic regimen were excluded from the study.
* Children 's parents who are smokers (passive smoking ) to reduce the confounding factors.
* No more than one child per family to be allowed into the study.
* Children who their parents refuse to participate in the study.

Ages: 7 Years to 14 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-09-20 (Estimated); Study Completion 2024-03-20 (Estimated)

PRIMARY OUTCOMES:
The incidence of patient with mild to moderate gingivitis using international periodantal disease detection . | 3 weeks after mouth wash application
  The measure will be done using international detection and assessment criteria for diagnosing mild to moderate gingivitis by naked eye and periodantal probe.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Yousif, Principal Investigator — University of Baghdad
Locations (1):
- the specialist dental center in Diyala city, Baghdad, Iraq